CLINICAL TRIAL: NCT06067919
Title: Assessment of the Applicability and Acceptability of an Algorithm to Guide the Prescription of 1st and 2nd Generation Cephalosporins as Part of Intraoperative Antibiotic Prophylaxis in Patients With a Declared Allergy to Penicillin
Acronym: PROPHYLAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: APHP220837
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-05

CONDITIONS: Adult Patients Who Declare an Allergy to Penicillin During Anaesthetic Consultation Without Any Allergy Work up That Could Confirm This Declaration; Good Comprehension of French Language
MeSH Terms: interventions — Decision Trees

STUDY DESIGN:
Intervention Model Description: assess the impact of disseminating of a decision tree on prescribing practices, a cluster randomised, stepped-wedge, multicentre, national, interventional, pragmatic and open study will be carried out.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- usual care (No Intervention)
- use of a decision tree to guide antibiotic prophylaxis prescription (Experimental)
  Interventions: Other: decision tree for the choice of intraoperative antibiotic prophylaxis

INTERVENTIONS:
Other: decision tree for the choice of intraoperative antibiotic prophylaxis — Presentation of a decision tree to anaesthetists to guide the choice of intraoperative antibiotic prophylaxis
  Arms: use of a decision tree to guide antibiotic prophylaxis prescription

SUMMARY:
According to the Centers for Disease Control and Prevention (CDC), a surgical site infection (SSI) is an infection that occurs after surgery at the site where the surgery was performed. The prevalence of SSIs is difficult to obtain and is probably underestimated, as many SSIs occur after the patient has been discharged from hospital and are not taken into account. SSIs are responsible for an increase in length of stay, mortality and costs. Their prevention is therefore essential in the operating theater, and has been the subject of recommendations recently updated by the CDC. The first line of prevention is the administration of prophylaxis antibiotic adapted to the surgical procedure, administered within a specific timeframe in order to achieve an effective bactericidal concentration in the tissues at the time of the surgical incision. In France, in the United States and for the WHO, the recommended first line of antibiotic prophylaxis is most often an agent from the beta-lactam family, a penicillin or a cephalosporin, with the exception of ophthalmological surgery. No strategy is described for the management of patients with a reported allergy to penicillin, apart from the recommendation of therapeutic alternatives.

The use of a decision-making strategy in the operating theater for patients with a reported allergy to penicillin therefore appears necessary and is recommended by experts. In the intraoperative context, the application of a strategy would make it possible to guide the use of cephalosporins, without removing the "penicillin allergy" label from the patient, but by proposing an alternative via the use of a cephalosporin depending on the probability of the risk of a real allergy to penicillin, according to the description of the former reaction.

DETAILED DESCRIPTION:
According to the Centers for Disease Control and Prevention (CDC), a surgical site infection (SSI) is an infection that occurs after surgery at the site where the surgery was performed. The prevalence of SSIs is difficult to obtain and is probably underestimated, as many SSIs occur after the patient has been discharged from hospital and are not taken into account. SSIs are responsible for an increase in length of stay, mortality and costs. Their prevention is therefore essential in the operating theater, and has been the subject of recommendations recently updated by the CDC. The first line of prevention is the administration of prophylaxis antibiotic adapted to the surgical procedure, administered within a specific timeframe in order to achieve an effective bactericidal concentration in the tissues at the time of the surgical incision. In France, in the United States and for the WHO, the recommended first line of antibiotic prophylaxis is most often an agent from the beta-lactam family, a penicillin or a cephalosporin, with the exception of ophthalmological surgery. No strategy is described for the management of patients with a reported allergy to penicillin, apart from the recommendation of therapeutic alternatives.

The use of a decision-making strategy in the operating theater for patients with a reported allergy to penicillin therefore appears necessary and is recommended by experts. In the intraoperative context, the application of a strategy would make it possible to guide the use of cephalosporins, without removing the "penicillin allergy" label from the patient, but by proposing an alternative via the use of a cephalosporin depending on the probability of the risk of a real allergy to penicillin, according to the description of the former reaction.

The main objective is to assess the impact on first and second generation cephalosporins prescription rate of a decision tree designed to guide the prescription of first and second generation cephalosporins in patients with a self-reported allergy to penicillin.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years;
* Patients with a good French understanding
* Who declare themselves allergic to penicillin and who have not benefit from an allergy work-up to explore their allergies and possible therapeutic alternatives;
* Requiring antibiotic prophylaxis with either first or second generation cephalosporins for elective or emergency surgery.

Exclusion Criteria:

* Refusal to sign informed consent
* Patient under legal protection ;
* Pregnant women;
* Patient scheduled for surgery requiring first-line antibiotic prophylaxis with an agent other than first and second generation cephalosporins (such as amoxicillin/clavulanate or vancomycin) according to the recommendations of the French Society of Anaesthesia and Intensive Care (SFAR) in one of the investigating centres;
* Patient declaring an allergy to antibiotics other than penicillins.
* Not affiliated to a social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
prescription of 1st generation cephalosporins | surgery day
  Rate of prescription of 1st cephalosporins for intraoperative antibiotic prophylaxis.
prescription of 2nd generation cephalosporins | surgery day
  Rate of prescription of 2nd generation cephalosporins for intraoperative antibiotic prophylaxis.

SECONDARY OUTCOMES:
surgical site infections (SSI) | 30 days after surgery
  number of surgical site infections (SSI)
new surgery due to surgical site infections (SSI) | 30 days after surgery
  number of new surgery due to SSI
intraoperative hypersensitivity reactions attributable to antibiotic prophylaxis | surgery day
  Number of intraoperative hypersensitivity reactions attributable to antibiotic prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Mouna Ben Rehouma, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bichat hospital, Paris, France